CLINICAL TRIAL: NCT02370823
Title: A Controlled Surveillance of the Osteoarthritic Knee Microenvironment With Regenexx® SD Treatment
Status: Terminated | Type: Observational
Why Stopped: Terminated early for poor study design.
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RSI2014-LAB01
Record Dates: First submitted 2015-02-10; First posted 2015-02-25 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Synovial Fluid an QC bone marrow sample may be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee OA Treated with Regenexx SD: 20 subjects with unilateral knee osteoarthritis. Collection of synovial fluid from both knees will serve as the experimental condition, i.e. the osteoarthritic knee, and the matched control, i.e. the knee not demonstrating signs of osteoarthritis. Alterations in the concentration of the synovial fluid proteins and cellular components will be evaluated up to 6 weeks post-Regenexx® SD - Same Day Bone Marrow Concentrate Injection treatment.
  Interventions: Procedure: Regenexx SD

INTERVENTIONS:
Procedure: Regenexx SD — stem cell treatment
  Other Names: Bone Marrow Concentrate

SUMMARY:
The primary objective of this study is to determine the levels of proteins and/or cellular components of the synovial fluid that are indicative of microenvironment phenotypes of the osteoarthritic knee compared to unilateral unaffected joints pre-injection to 6 weeks post-Regenexx® SD treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the levels of proteins and/or cellular components of the synovial fluid that are indicative of microenvironment phenotypes of the osteoarthritic knee compared to unilateral unaffected joints pre-injection to 6 weeks post-Regenexx SD treatment (day 0).

Secondary objective is an evaluation of possible direct and/or indirect associations between the measured levels of proteins and/or cellular components of the synovial fluid in the osteoarthritic knee joint with the administration of the Regenexx SD treatment. The secondary objective will include MRI evidence of cartilage repair; incidence of post-operative complications, adverse events, re-injections, and surgical intervention; change in pain score and use of pain medications.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the IRB approved Informed Consent
2. Unilateral osteoarthritic male or female ages 35-85
3. Pain, swelling, and/or functional disability in the affected knee consistent with osteoarthritis in one knee joint
4. Physical examination consistent with osteoarthritis in one knee joint
5. Restricted range of motion of the affected knee (<135 degrees in flexion and/or >0 degrees of extension)
6. Kellgren-Lawrence grade 2 or greater knee osteoarthritis with diagnostic MR imaging of the affected knee showing osteoarthritis
7. Limited knee effusion in osteoarthritic knee (i.e. not more than 20 ml of visible joint fluid on ultrasound examination of the knee.)
8. Normal range of motion of the unaffected knee
9. No sign of pain, swelling, and/or functional disability of the unaffected knee
10. No history of acute injury in the unaffected knee
11. Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion Criteria:

1. Knee injections of any type within 6 months prior to the study.
2. Inflammatory or auto-immune based joint diseases or other lower extremity pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
3. Quinolone or Statin induced myopathy/tendinopathy
4. Symptomatic lumbar spine pathology (e.g. radicular pain)
5. Severe neurogenic inflammation of the cutaneous nerves about the knee or thigh (i.e. evidence of complex regional pain syndrome or central sensitization with allodynia present on exam).
6. Contraindications for MRI
7. Tested positive or has been treated for a malignancy in the past five years or is suspected of having a malignancy or is currently undergoing radiation or chemotherapy treatment for a malignancy anywhere in the body, whether adjacent to or distant from the proposed injection site
8. Condition represents a worker's compensation case
9. Currently involved in a health-related litigation procedure
10. Is pregnant
11. Bleeding disorders
12. Currently taking anticoagulant or immunosuppressive medication
13. Allergy or intolerance to study medication
14. Use of chronic opioid
15. Documented history of drug abuse within six months of treatment

18) Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will have unilateral knee OA as evidenced with physical examination and MRI. Subjects will be recruited from the physician practice and will be males and females age 35-85.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Median change in protein concentration or percentage of cellular subpopulations | 6 weeks compared to baseline
  A comparison of the patient temporal median change in protein concentration or percentage of cellular subpopulations from pre-injection to 6 weeks post- Regenexx SD treatment.

SECONDARY OUTCOMES:
Mean Change in Pain Scale from baseline to 6 weeks | 6 weeks
  Mean Numeric Pain Scale
Mean Change in IKDC Scores from baseline to 6 weeks | 6 weeks
  Mean Patient Reported Pain and Function Scale
Incidence and time to resolution of post-operative complications and adverse events | 6 weeks
  Incidence and time to resolution of post-operative complications and adverse events
Incidence and time to re-injection/re-operation | 6 weeks
  Incidence and time to re-injection/re-operation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No